CLINICAL TRIAL: NCT04190147
Title: Ocular Morphology and Visual Function in Relation to Growth, Metabolic, Cardiovascular, and Neuropsychiatric Status, and Quality of Life in Adolescents Born Moderate-to-late Preterm
Brief Title: Eye and Growth in Adolescents Born Moderate-to-late Preterm
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: MLP15
Record Dates: First submitted 2019-08-22; First posted 2019-12-09 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-01

CONDITIONS: Preterm Birth; Visual Impairment; Eye Abnormalities
Keywords: Moderate-to-late preterm
MeSH Terms: conditions — Premature Birth; Vision Disorders; Eye Abnormalities | interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate-to-late preterm group
  Interventions: Other: Structural, functional and metabolic eye examinations
- Full-term group
  Interventions: Other: Structural, functional and metabolic eye examinations

INTERVENTIONS:
Other: Structural, functional and metabolic eye examinations — Structural, functional and metabolic eye examinations

SUMMARY:
During recent years, the interest in studying the risks of being born moderate-to-late preterm (MLP), defined as birth between gestational week 32 to 36, has increased. Today the investigators know that morbidity and mortality are significantly higher in these individuals compared to individuals born full-term. However, few studies have focused on the development of the eye in MLP individuals. The purpose of the study is to evaluate eye morphology and visual function in relation to growth, metabolism, blood pressure, neuropsychiatric factors, and quality of life in adolescents born MLP. The results of the examinations will be compared to an age-matched control group. The study will evaluate the structural, functional, and metabolic aspects of the eye with the hypothesis that early eye abnormalities may detect the risk of developing metabolic and cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Born moderate-to-late preterm.
* Born in Gothenburg, Sweden.
* Born between years 2002 and 2004.

Exclusion Criteria:

* Chromosomal abnormalities.
* Syndromes.
* Severe malformations.
* Asphyxia.
* Language difficulties.
* Psychosocial problems at birth.
* Severe maternal illness.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Year 2002 to 2004, 247 children born moderate-to-late preterm i Gothenburg, Sweden, were enrolled in a prospective, longitudinal and population-based cohort study. These children will be asked to participate in the present follow-up study 15 years later. The age-matched control group born full-term will be recruited from schools in Gothenburg.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Optic disc area. | Through study completion, an average of 6 months
  Optic disc area measured with Optical coherence tomography (OCT, Topcon).
Visual acuity. | Through study completion, an average of 6 months.
  Visual acuity measured with Early Treatment Diabetic Retinopathy Study (ETDRS) scores.
Blood pressure. | Through study completion, an average of 6 months.
  Systolic and diastolic blood pressure measured with blood pressure cuffs.
Blood concentration of Hemoglobin A1c (HbA1c). | Through study completion, an average of 6 months.
  Blood samples of HbA1c.
Autism Spectrum Screening Questionnaire (ASSQ). | Through study completion, an average of 6 months.
  The ASSQ consists of 27 items and is scored using a likert scale, with the following alternatives: "not true" (0 points), "somewhat true" (1 point) and "certainly true" (2 points).
Pediatric Quality of Life Inventory (PedsQL). | Through study completion, an average of 6 months.
  PedsQL is a questionnaire measuring health-related quality of life in children and adolescents aged 2 to 18 years. It consists of 23 items including physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). It has a 5-point response scale: "never a problem" (0 points), "almost never a problem" (1 point), "sometimes a problem" (2 points), "often a problem" (3 points), "almost always a problem" (4 points).
Weight. | Through study completion, an average of 6 months
  Weight measured in kilograms.
The Swanson, Nolan, and Pelham Rating Scale (SNAP-IV). | Through study completion, an average of 6 months.
  Screening questionnaire for attention deficit hyperactivity disorder (ADHD) consisting of 26 items rated on a 4-point scale: "not at all" (0 points), "just a little" (1 point), "quite a bit" (2 points) and "very much" (3 points).
Refraction. | Through study completion, an average of 6 months.
  Visual refraction measured with an autorefractor (Topcon).
Height. | Through study completion, an average of 6 months.
  Height measured in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of neuroscience and physiology, Gothenburg, Västra Götaland County, Sweden